CLINICAL TRIAL: NCT05185479
Title: Analysis of ADVerse evENTs in Anesthesia Using ARtificial IntelligencE
Acronym: ADVENTURE
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8505
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Allergic Reaction
Keywords: Allergic Reaction; Adverse events; Health database; Natural Language Processing
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The interest of health databases in anesthesia is no longer to be demonstrated. The aim of this research was to develop a natural language processing approach to establish a classification of adverse events observed during the perioperative period and to facilitate their analysis:

The main objective of the study was to identify what a "naïve" unsupervised model would discover based on Adverse Event (AE) descriptions. Our second goal was to identify apparently unrelated events whose combination could favor the occurrence of an AE

ELIGIBILITY:
Inclusion Criteria:

* Minors and adults having had an allergic reaction associated with care
* Having had an adverse event reported by an anesthetist between January 01, 2009 and June 30, 2020

Exclusion Criteria:

- Patient not meeting the inclusion criteria

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Minors and adults having had an allergic reaction associated with care, and having had an adverse event reported by an anesthetist between January 01, 2009 and June 30, 2020
Sampling Method: Non-Probability Sample
Enrollment: 9559 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Development of a natural language processing approach to establish a classification of adverse events observed during the perioperative period and to facilitate their analysis. | Files analysed retrospectively from January 01, 2009 to June 30, 2020 will be examined]
  The aim of this research was to develop a natural language processing approach to establish a classification of adverse events observed during the perioperative period and to facilitate their analysis:
  The main objective of the study was to identify what a "naïve" unsupervised model would discover based on Adverse Event (AE) descriptions. Our second goal was to identify apparently unrelated events whose combination could favor the occurrence of an AE

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Michel MERTES, MD, PhD, Principal Investigator — Service d'Anesthésie et Réanimation chirurgicale - CHU de Strasbourg - France
Locations (1):
- Service d'Anesthésie et Réanimation chirurgicale - CHU de Strasbourg - France, Strasbourg, France

REFERENCES:
- [Derived] Mertes PM, Morgand C, Barach P, Jurkolow G, Assmann KE, Dufetelle E, Susplugas V, Alauddin B, Yavordios PG, Tourres J, Dumeix JM, Capdevila X. Validation of a natural language processing algorithm using national reporting data to improve identification of anesthesia-related ADVerse evENTs: The "ADVENTURE" study. Anaesth Crit Care Pain Med. 2024 Aug;43(4):101390. doi: 10.1016/j.accpm.2024.101390. Epub 2024 May 6. PMID 38718923